CLINICAL TRIAL: NCT02451852
Title: A Multi-center, AZD9291 Expanded Access Program for the Treatment of Patients With Advanced/Metastatic EGFR T790M Mutation-positive Non-small Cell Lung Cancer (NSCLC) Who Have Received Prior EGFR TKI Therapy
Brief Title: AZD9291 US Expanded Access Program
Status: No longer available | Type: Expanded Access
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5160C00021
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: EGFR T790M Mutation Positive NSCLC
MeSH Terms: interventions — osimertinib

INTERVENTIONS:
Drug: AZD9291 — AZD9291 80mg tablet once daily, open label

SUMMARY:
To provide access to AZD9291 for adult patients with advanced/metastatic, epidermal growth factor receptor T790M mutation-positive non-small cell lung cancer.

DETAILED DESCRIPTION:
- This is a multi-center, AZD9291 expanded access protocol for the treatment of adult patients with advanced/metastatic EGFR T790M mutation-positive non-small cell lung cancer (NSCLC) who have received prior EGFR TKI therapy and at least one additional line of therapy (≥ 3rd line). Local testing is accepted for confirmation of T790 mutation status. Eligible patients will be enrolled to receive AZD9291 (80mg orally, once daily) for as long as the access program remains open and they are continuing to show clinical benefit, as judged by the treating physician

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any treatment protocol-specific procedures
* Patients aged at least 18 years
* Locally advanced or metastatic EGFRm NSCLC, not amenable to curative surgery or radiotherapy with confirmation of the presence of the T790M mutation
* Two lines of prior therapy including at least one EGFR TKI
* World Health Organization (WHO) performance status 0-2.
* Females of child-bearing potential must use adequate contraceptive measures, not be breast-feeding and have negative pregnancy test prior to start of dosing.
* Males patients should be willing to use barrier contraception.

Exclusion Criteria:

* Previous treatment with AZD9291
* Patients currently receiving (or unable to stop use at least 1 week prior to receiving the first dose of AZD9291) any treatment known to be potent inhibitors or inducers of CYP3A4
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, or significantly impaired bone marrow reserve or organ function, including hepatic and renal impairment, which in the clinician's opinion would significantly alter the risk/benefit balance, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV).
* Patients with symptomatic CNS metastases who are neurologically unstable
* Past medical history of ILD, drug-induced ILD, radiation pneumonitis requiring steroid treatment, or any evidence of clinically active ILD
* Any of the following cardiac criteria:

  1. Mean resting corrected QT interval (QTc using Fredericia's formula) > 470 msec
  2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block, second degree heart block)
  3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval
* Any unresolved toxicity from prior therapy Common Terminology Criteria for Adverse Events (CTCAE) > grade 3 at the time of starting treatment in the access program
* History of hypersensitivity to AZD9291 (or drugs with a similar chemical structure or class to AZD9291) or any excipients of these agents
* Males and females of reproductive potential who are not using an effective method of birth control and females who are pregnant or breastfeeding or have a positive (urine or serum) pregnancy test prior to access program entry

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Research Site, Anaheim, California
  - Research Site, Beverly Hills, California
  - Research Site, Burbank, California
  - Research Site, Santa Barbara, California
  - Research Site, Santa Rosa, California
  - Research Site, Manchester, Connecticut
  - Research Site, Boca Raton, Florida
  - Research Site, Fleming Island, Florida
  - Research Site, Athens, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Chicago, Illinois
  - Research Site, Chevy Chase, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Lincoln, Nebraska
  - Research Site, Paramus, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, Fresh Meadows, New York
  - Research Site, Mineola, New York
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Warrenton, Virginia
  - Research Site, Lacey, Washington
  - Research Site, Seattle, Washington